CLINICAL TRIAL: NCT03931850
Title: Does Neurostimulation Improve Efficacy for Ultrasound-Guided Transperineal Pudendal Nerve Block In Children: A Randomized Clinical Trial
Brief Title: Does Neurostimulation Improve Efficacy for Ultrasound-Guided Transperineal Pudendal Nerve Block In Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ramathibodi Hospital (Other)
Collaborators: Maharaj Nakorn Chiang Mai Hospital (Other)
Responsible Party: Principal Investigator, Witchaya Supaopaspan, Principal investigator, Ramathibodi Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12-61-49
Record Dates: First submitted 2019-04-23; First posted 2019-04-30 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Phimosis
Keywords: Pudendal nerve; circumcision; pediatric
MeSH Terms: conditions — Phimosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual guidance (ultrasound and neurostimulation) (Experimental): This arm : patients will be received pudendal nerve block by dual guidance technique ( ultrasound and neurostimulation)
  Interventions: Procedure: Pudendal nerve block
- ultrasound-guided only (Active Comparator): This arm : patients will be received pudendal nerve block by ultrasound-guided only.
  Interventions: Procedure: Pudendal nerve block

INTERVENTIONS:
Procedure: Pudendal nerve block — Pudendal nerve block is the one of peripheral nerve block. Injection local anesthetic medication around this nerve can provide analgesia around perineal area.

SUMMARY:
This study aim to compare efficacy of transperineal pudendal nerve block between 2 techniques, by dual guidance (ultrasound and neurostimulation) vs by ultrasound-guided only, in pediatric patients who undergo circumcision.

Primary outcome : Block efficacy will be assessed from ratio of patients who receive opioids in immediate postoperative period.

Secondary outcomes :

* This study also measure other aspects of pain which can reflect the block efficacy including pain score in 24 hours, postoperative analgesic requirement in 24 hours, time to first analgesia, block success rate.
* Block performance : imaging time, needling time, total performance time,
* Block safety : collect complications from block including vascular/rectal puncture, bleeding (hematoma), local anesthetic systemic toxicity, voiding difficulty
* Parental satisfaction will be also collected which scoring use 1-5 metric.

DETAILED DESCRIPTION:
Pain after circumcision is moderate to high level. Inadequate pain control leads to severe agitation, swelling of the wound, neurobehavioral change, lower parental satisfaction. Pain control for circumcision including topical, Dorsal penile nerve block, Caudal block. Topical is inadequate to control post-circumcision pain. Dorsal penile nerve block is not completely cover every areas of penis and also has 4-6.7% failure rate. For Caudal block provides good pain control but it is not proper for ambulatory surgery because of common adverse effects such as motor weakness, urinary retension, moreover it has short duration only 6 hours after block.

In the last 15 years, large-scale studies from many countries studied the safety of regional anesthesia in pediatric patients. It was found that the central neuraxial and peripheral nerve blockage can be done safely, especially using ultrasound-guided to increase safety. Therefore, regional anesthesia is extensive performed in pediatric patients with the main purpose of controlling postoperative pain after surgery, reducing the use of opioids analgesics which may cause respiratory depression, especially in young children.Pudendal nerve block for postoperative pain relief for circumcision, hypospadias has been shown to be effective.

Pudendal nerve derives from anterior rami of spinal nerve root S2-S4 then runs into Alcock's canal and enters the ischiorectal fossa. In this area, pudendal nerve will separate to 3 branches 1) Dorsal penile nerve 2) Perineal branch 3) Rectal branch, therefore pudendal nerve block can provide effective postoperative pain control for surgery around perineal area such as circumcision, hypospadias, anoplasty.

There were several studies on the effectiveness of pudendal nerve block for treating pudendal neuralgia and to control pain after hemorrhoidectomy in adult patients. For pediatric patients, the effectiveness of pudendal nerve block in circumcision surgery compared to the dorsal nerve block was found that in the group receiving the pudendal nerve block, the pain score is lower, with less painkiller and longer pain control. In addition, the study of the pudendal nerve block in pediatric patients who underwent hypospadias in comparison to caudal block, the group that received the pudendal nerve block had a longer duration of pain relief.It can be concluded that the pudendal nerve block is more effective in pain control than the traditional dorsal penile nerve block for circumcision and more effective than caudal block for hypospadias. In addition, it can avoid side effects from caudal block, such as motor weakness, urinary retension, and can be a good alternative pain relief for patients who have contraindication to neuraxial block.

However, the effectiveness of pain control by the pudendal nerve block method is also different, which may be the technical difference of the block. In principle, for the performing peripheral nerve block, the more injection of local anesthetics approach the nerve, the more efficacy will also be followed, and the duration of action will be longer. But the injection near the nerve will increase the chance of causing nerve damage.Therefore, the ideal method of the peripheral nerve block is to inject as close to the nerve as possible without causing injury to the nerves, which is currently a device that can be used to identify the position of the nerve. 1) Using Nerve Stimulator (NS), stimulator by looking at the response of muscles when electrically stimulated, the position used to identify the proximity of the needles to the nerve is the response of the muscle at 0.5 milliampere and no response when using electricity 0.2 milliampere,which indicates that the needle tip is in the right position, not too close or too far 2) Using an ultrasound-guided, which allows to see the position of nerves, blood vessels, and adjacent organs, which can be injected at the point without harm. 3) Using dual-guidance (both ultrasound together with nerve stimulator, which is expected to benefit both of these methods.

The study conducted by Naja and Kendigelen supported that the use of the Nerve Stimulator-guided could provide 100% success rate with patients requiring extra painkillers within the first 24 hours only 7.5-20%. The performance time of block is 2-8 minutes. Later, the study by Gaudet-Ferrand that performed pudendal nerve block under U/S-guided only in pediatric patients who underwent perineum surgery, they reported the success rate only 88% and 60% of patients required opioids in recovery room. Which , compared to previous studies, there was no patient who wanted opioid in recovery room.That show the use of U/S guided pudendal nerve block only is less effective than performing by Nerve Stimulator-guided, which possible cause is U/S could not identify pudendal nerve in every patients.That makes the injection too far from nerve or can injure the nerve unintentionally.

However, using only the Nerve Stimulator still has a risk of injury to important organs such as rectum or adjacent vessels, especially in small children or performing by less expertise. So using U/S will increase safety of block.

This study will find out the effectiveness of performing transperineal pudendal nerve block by dual guidance which use both of NS and U/S guided compare with using U/S guided only. Assuming that the dual guidance technique should increase the effectiveness of the pudendal nerve block compare to the use of U/S guided alone. The primary outcome is the efficacy of postoperative pain control by evaluating the proportion of patients who need opioids during immediate postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* Age between 8 months to 7 years
* American Society of Anesthesiologists (ASA) class 1-3
* Undergoing elective circumcision
* Consent to participate in research by the parents signing the letter of intent to participate in the research project

Exclusion Criteria:

* Refuse to receive regional nerve block
* Allergic to Bupivacaine or Paracetamol
* Coagulopathy
* Severe coexisting liver or kidney disease
* There is a wound or infection in the pelvis area
* Underlying neurodeficit including attention deficit, cerebral palsy, Down's syndrome
* Parents cannot evaluate pain scores
* Patients or parents have willing to withdraw from research.

Ages: 8 Months to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2019-04-30 (Actual); Primary Completion 2020-07-10 (Estimated); Study Completion 2020-07-10 (Estimated)

PRIMARY OUTCOMES:
the proportion of patients who need opioids in recovery room | 1 hour (in recovery room)
  the proportion of patients who need opioids in recovery room in each group

SECONDARY OUTCOMES:
Block success rate | Intraoperation
  No increasing of blood pressure or heart rate more than 10 % of baseline before incision
Postoperative analgesic requirement in 24 hours | 24 hours postoperation
  Postoperative analgesics including
  1. Fentanyl : unit is microgram
  2. paracetamol : milligrams
Time to first analgesic medication | 24 hours after operation
  Time (in hours) that patients received the first analgesic medications.
Pain score will be assessed by Face Legs Activity Cry Consolability scale (FLACCs) | 6 hours after arriving the ward
  use Face Legs Activity Cry Consolability scale patients will be assessed by FLACCs , 6 times
  * In recovery room : will assess every 15 minutes, 4 times
  * Time at Arriving the ward
  * 6 hours after arriving the ward
  FLACC score (score 1-10, minimum is 1, maximum is 10) FLACC score >3 , patients will be received fentanyl 0.5 micrograms/kilogram
Parents' Postoperative Pain Measure-Short Form (PPPM-SF) | 6 hours after arriving the ward untill 24 hours after operation
  Patients will be assessed by PPPM-SF by parents every 6 hours PPPM-SF (score 1-10, minimum is 1, maximum is 10) score > 1 , patients will be received paracetamol 15 milligrams/ kilogram
Performance time | Intraoperation
  Time spent for performing pudendal nerve block ( minutes)
Complications from pudendal nerve block | 24 hours after operation
  incidence of :
  * vaacular puncture
  * rectal puncture
  * internal organ injury
  * local anesthetic toxicity
  * voiding difficulty
Parental satisfaction score | 24 hours after operation
  Parental satisfaction score : scoring from 1-5 ( 1 = unsatisfied, 5=the most satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Witchaya Supaopaspan, medical, Principal Investigator — Ramathibodi Hospital; Artid Samerchua, medical, Study Director — Maharaj Nakorn Chiang Mai Hospital
Locations (1):
- Ramathibodi Hospital, Bangkok, Ratchathewi, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yeoman PM, Cooke R, Hain WR. Penile block for circumcision? A comparison with caudal blockade. Anaesthesia. 1983 Sep;38(9):862-6. doi: 10.1111/j.1365-2044.1983.tb12251.x. PMID 6625133
- [Background] Vater M, Wandless J. Caudal or dorsal nerve block? A comparison of two local anaesthetic techniques for postoperative analgesia following day case circumcision. Acta Anaesthesiol Scand. 1985 Feb;29(2):175-9. doi: 10.1111/j.1399-6576.1985.tb02180.x. PMID 3976329
- [Background] Tree-Trakarn T, Pirayavaraporn S. Postoperative pain relief for circumcision in children: comparison among morphine, nerve block, and topical analgesia. Anesthesiology. 1985 Apr;62(4):519-22. doi: 10.1097/00000542-198504000-00027. No abstract available. PMID 3885795
- [Background] Walker BJ, Long JB, Sathyamoorthy M, Birstler J, Wolf C, Bosenberg AT, Flack SH, Krane EJ, Sethna NF, Suresh S, Taenzer AH, Polaner DM, Martin L, Anderson C, Sunder R, Adams T, Martin L, Pankovich M, Sawardekar A, Birmingham P, Marcelino R, Ramarmurthi RJ, Szmuk P, Ungar GK, Lozano S, Boretsky K, Jain R, Matuszczak M, Petersen TR, Dillow J, Power R, Nguyen K, Lee BH, Chan L, Pineda J, Hutchins J, Mendoza K, Spisak K, Shah A, DelPizzo K, Dong N, Yalamanchili V, Venable C, Williams CA, Chaudahari R, Ohkawa S, Usljebrka H, Bhalla T, Vanzillotta PP, Apiliogullari S, Franklin AD, Ando A, Pestieau SR, Wright C, Rosenbloom J, Anderson T; Pediatric Regional Anesthesia Network Investigators. Complications in Pediatric Regional Anesthesia: An Analysis of More than 100,000 Blocks from the Pediatric Regional Anesthesia Network. Anesthesiology. 2018 Oct;129(4):721-732. doi: 10.1097/ALN.0000000000002372. PMID 30074928
- [Background] Ivani G, Suresh S, Ecoffey C, Bosenberg A, Lonnqvist PA, Krane E, Veyckemans F, Polaner DM, Van de Velde M, Neal JM. The European Society of Regional Anaesthesia and Pain Therapy and the American Society of Regional Anesthesia and Pain Medicine Joint Committee Practice Advisory on Controversial Topics in Pediatric Regional Anesthesia. Reg Anesth Pain Med. 2015 Sep-Oct;40(5):526-32. doi: 10.1097/AAP.0000000000000280. PMID 26192549
- [Background] Suresh S, Ecoffey C, Bosenberg A, Lonnqvist PA, de Oliveira GS Jr, de Leon Casasola O, de Andres J, Ivani G. The European Society of Regional Anaesthesia and Pain Therapy/American Society of Regional Anesthesia and Pain Medicine Recommendations on Local Anesthetics and Adjuvants Dosage in Pediatric Regional Anesthesia. Reg Anesth Pain Med. 2018 Feb;43(2):211-216. doi: 10.1097/AAP.0000000000000702. PMID 29319604
- [Background] Tutuncu AC, Kendigelen P, Ashyyeralyeva G, Altintas F, Emre S, Ozcan R, Kaya G. Pudendal Nerve Block Versus Penile Nerve Block in Children Undergoing Circumcision. Urol J. 2018 May 3;15(3):109-115. doi: 10.22037/uj.v0i0.4292. PMID 29299888
- [Background] Kendigelen P, Tutuncu AC, Emre S, Altindas F, Kaya G. Pudendal Versus Caudal Block in Children Undergoing Hypospadias Surgery: A Randomized Controlled Trial. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):610-5. doi: 10.1097/AAP.0000000000000447. PMID 27501015
- [Background] Naja ZM, Ziade FM, Kamel R, El-Kayali S, Daoud N, El-Rajab MA. The effectiveness of pudendal nerve block versus caudal block anesthesia for hypospadias in children. Anesth Analg. 2013 Dec;117(6):1401-7. doi: 10.1213/ANE.0b013e3182a8ee52. PMID 24257391
- [Background] Naja Z, Al-Tannir MA, Faysal W, Daoud N, Ziade F, El-Rajab M. A comparison of pudendal block vs dorsal penile nerve block for circumcision in children: a randomised controlled trial. Anaesthesia. 2011 Sep;66(9):802-7. doi: 10.1111/j.1365-2044.2011.06753.x. Epub 2011 Jul 25. PMID 21790518
- [Background] Gaudet-Ferrand I, De La Arena P, Bringuier S, Raux O, Hertz L, Kalfa N, Sola C, Dadure C. Ultrasound-guided pudendal nerve block in children: A new technique of ultrasound-guided transperineal approach. Paediatr Anaesth. 2018 Jan;28(1):53-58. doi: 10.1111/pan.13286. Epub 2017 Dec 5. PMID 29205687
- [Background] Hecht S, Pineda J, Bayne A. Ultrasound-guided Pudendal Block Is a Viable Alternative to Caudal Block for Hypospadias Surgery: A Single-Surgeon Pilot Study. Urology. 2018 Mar;113:192-196. doi: 10.1016/j.urology.2017.11.006. Epub 2017 Nov 16. PMID 29155191
- [Background] Mamlouk MD, vanSonnenberg E, Dehkharghani S. CT-guided nerve block for pudendal neuralgia: diagnostic and therapeutic implications. AJR Am J Roentgenol. 2014 Jul;203(1):196-200. doi: 10.2214/AJR.13.11346. PMID 24951215
- [Background] Naja Z, Ziade MF, Lonnqvist PA. Nerve stimulator guided pudendal nerve block decreases posthemorrhoidectomy pain. Can J Anaesth. 2005 Jan;52(1):62-8. doi: 10.1007/BF03018582. PMID 15625258
- [Background] Naja Z, El-Rajab M, Al-Tannir M, Ziade F, Zbibo R, Oweidat M, Lonnqvist PA. Nerve stimulator guided pudendal nerve block versus general anesthesia for hemorrhoidectomy. Can J Anaesth. 2006 Jun;53(6):579-85. doi: 10.1007/BF03021848. PMID 16738292
- [Background] Chow S, Shao J, Wang H. Sample Size Calculations in Clinical Research. 2nd ed: Chapman&Hall/CRC; 2003